CLINICAL TRIAL: NCT04104750
Title: The Assessment of Fatigue and Quality of Life in Patients With Bone Tumor, Undergoing Chemotherapy Treatment and Possible Predictive Factors
Brief Title: The Assessment of Fatigue and Quality of Life in Patients With Bone Tumor,
Acronym: Fatigue-ONCO
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: Fatigue-ONCO
Record Dates: First submitted 2019-09-18; First posted 2019-09-26 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Fatigue Syndrome, Chronic; Bone Tumor; Quality of Life
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Bone Neoplasms | interventions — TES

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment scales (BFI, QLQ, TESS) — the patient's Fatigue will be measured during the treatment period with antiblastic drugs and part of the followup period. To this end the BFI scale validated in Italian will be used (Mendoza et al 1999; Catania et al, 2013) which includes 9 items with a score for each of 0 to 10 and a consequent total score from 0 to 90. The measurement will take place in 4 times: the day of enrollment, 6 months, 12 months and 24 months after enrollment.the quality of life of patients measured by the EORTC QLQ C-30 scale (Aaronson et al, 1993) and the level of autonomy measured by the TESS scale (Davis et al, 1996) in 4 steps: the enrollment day , at 6 months, at 12 months and at 24 months from enrollment.

SUMMARY:
The aim of the present observational study is to evaluate and describe the evolution over time of the fatigue and the quality of life of patients with bone tumor, in Rizzoli Orthopedic Institute, Chemotherapy ward, during the chemotherapy treatment and in the first phase of follow-up and to identify possible prognostic factors. Such knowledge is a necessary precondition for identifying patients and the periods most at risk due to the onset of fatigue, so as to be able to hypothesize adequate containment strategies.

DETAILED DESCRIPTION:
Fatigue syndrome It is a clinical condition, linked to the oncological pathology, extremely widespread and in patients undergoing chemotherapy and / or radiotherapy it is common in 80% of patients. Literature stress the need for systematic studies in cancer populations with different types of cancer and at different stages of the disease using patient-oriented fatigue assessment tools. The Brief Fatigue Inventory (BFI) is one of the scales used precisely in the evaluation of this syndrome and has proved to be a reliable and easy to use tool, also validated in Italian. Several authors have also shown that reduced physical activity and a worse quality of life are associated with fatigue, particularly in young patients.Several authors describe the experience of 11 new sarcoma patients undergoing chemotherapy treatment. Fatigue had been described as the prevalent symptom and was related to a worse quality of life.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with bone tumors who start a new chemotherapy treatment protocol

Exclusion Criteria:

* patients with little knowledge of the Italian language

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: all patients belonging to the Chemotherapy ward will be recruited consecutively for a new antiblastic treatment protocol. The process of informing and collecting the participants' consent will take place during the first admission in which intravenous administration of the chemotherapy will be started
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
the patient's Fatigue | through study completion, an average of 5years
  will be measured during the treatment period with antiblastic drugs and part of the followup period. To this end the Brief Fatigue Inventory scale validated in Italian will be used which includes 9 items with a score for each of 0 to 10 and a consequent total score from 0 to 90.

SECONDARY OUTCOMES:
the quality of life of patients | through study completion, an average of 5years
  Quality of life of patients measured by the European Organisation for Research and Treatment of Cancer quality of life scale

CONTACTS AND LOCATIONS:
Locations (1):
- Paola Coluccino, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Result] Catania G, Bell C, Ottonelli S, Marchetti M, Bryce J, Grossi A, Costantini M. Cancer-related fatigue in Italian cancer patients: validation of the Italian version of the Brief Fatigue Inventory (BFI). Support Care Cancer. 2013 Feb;21(2):413-9. doi: 10.1007/s00520-012-1539-z. Epub 2012 Jul 13. PMID 22790224
- [Derived] Morri M, Boccomino R, Brruku E, Romagnoli E, Boschi R, Raucci G, Bellina Terra A, Coluccino P. Fatigue, functional ability and quality of life in patients with bone and soft tissue sarcomas undergoing chemotherapy treatment: An observational study. Eur J Oncol Nurs. 2025 Feb;74:102736. doi: 10.1016/j.ejon.2024.102736. Epub 2024 Nov 16. PMID 39577033

DOCUMENTS (1):
  • Study Protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT04104750/Prot_000.pdf